CLINICAL TRIAL: NCT02181530
Title: Retrospective Data Collection Study in Patients With Macular Oedema Receiving OZURDEX®
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/OPH/RET/016
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Results first posted 2015-05-25 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Macular Edema; Retinal Vein Occlusion
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OZURDEX®: Retrospective data collection study of OZURDEX® (dexamethasone intravitreal implant 0.7 mg) administered at least once in accordance with routine clinical practice. No treatment (intervention) is administered as part of this study.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No treatment (intervention) is being administered as part of this study.

SUMMARY:
This study will use retrospective data to evaluate the safety and efficacy of OZURDEX® (dexamethasone intravitreal implant 0.7 mg) in the treatment of macular oedema due to retinal vein occlusion (RVO) in clinical practice. No intervention will be administered as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Macular oedema in at least one eye due to branch retinal vein occlusion (BRVO) or central vein occlusion (CRVO)
* Received at least one injection of OZURDEX® in the study eye

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with branch retinal vein occlusion (BRVO) or central retinal vein occlusion (CRVO) who received OZURDEX® as part of routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Warsaw, Poland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OZURDEX®
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | OZURDEX®
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.02 (13.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) in the Study Eye
Description: BCVA is measured in the study eye following each injection of OZURDEX® using a special eye chart. The number of letters read correctly Snellen fraction are converted to a decimal scale. There are 11 lines on a standard Snellen chart ranging from 0.1 (20/200) at worst to 2.0 (20/10) at best. 20/20 on the decimal scale is equal to 1.0. The lower the number of letters read correctly on the eye chart (lower number on the decimal scale) the worse the vision (or visual acuity). The higher the number of letters read correctly (higher number on the decimal scale), the better the vision (or visual acuity). A positive number improvement in the number of letters read means that the vision has improved.
Time Frame: Baseline, 7 to 12 weeks following the first OZURDEX® injection
Population: All participants with data available at the time-point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OZURDEX®
Number analyzed (Participants) | 43
units on a scale
  Baseline | 0.22 (0.22)
  Change from Baseline at 7 to 12 weeks (n=27) | 0.18 (0.25)

2. Secondary Outcome: Percentage of Patients With an Increase of 2 Lines or More in BCVA in the Study Eye
Description: BCVA following the injection of OZURDEX® is measured in the study eye using a special eye chart. BCVA measurements expressed in Snellen fractions were converted to logMAR units and approximate Early Treatment Diabetic Retinopathy Study (ETDRS) letter scores based on the formula: approximate ETDRS letters = 85 + 50 x log10 (Snellen fraction). The converted scores hereinafter are referred to as "approxETDRS letters" to distinguish the scores from visual acuity measurements obtained using the ETDRS chart. It was assumed that one line equals five ETDRS points. An increase of 2 lines or more indicates an improvement.
Time Frame: Baseline, Up to 17 Months
Population: All participants.
Measure: Number; unit: percentage of participants
Arm/Group | OZURDEX®
Number analyzed (Participants) | 43
percentage of participants | 63

3. Secondary Outcome: Percentage of Patients With an Increase of 3 Lines or More in BCVA in the Study Eye
Description: BCVA following the injection of OZURDEX® is measured in the study eye using a special eye chart. BCVA measurements expressed in Snellen fractions were converted to logMAR units and approximate ETDRS letter scores based on the formula: approximate ETDRS letters = 85 + 50 x log10 (Snellen fraction). The converted scores hereinafter are referred to as "approxETDRS letters" to distinguish the scores from visual acuity measurements obtained using the ETDRS chart. It was assumed that one line equals five ETDRS points. An increase of 3 lines or more indicates an improvement.
Time Frame: Baseline, Up to 17 Months
Population: All participants.
Measure: Number; unit: percentage of participants
Arm/Group | OZURDEX®
Number analyzed (Participants) | 43
percentage of participants | 53

4. Secondary Outcome: Change From Baseline in Retinal Thickness as Measured by Optical Coherence Tomography (OCT)
Description: OCT is measured in the study eye following each injection of OZURDEX®. OCT is a laser based non-invasive diagnostic system providing high-resolution imaging sections of the retina to assess retinal thickness. A negative change indicates an improvement
Time Frame: Baseline, 7 to 12 weeks following the first OZURDEX® injection
Population: All participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | OZURDEX®
Number analyzed (Participants) | 43
μm
  Baseline | 695.12 (212.71)
  Change from Baseline at 7 to 12 weeks (n=26) | -355.08 (184.72)

5. Secondary Outcome: Time to Improvement of 2 Lines or More in BCVA in the Study Eye
Description: BCVA following the injection of OZURDEX® is measured in the study eye using a special eye chart. BCVA measurements expressed in Snellen fractions were converted to logMAR units and approximate ETDRS letter scores based on the formula: approximate ETDRS letters = 85 + 50 x log10 (Snellen fraction). The converted scores hereinafter are referred to as "approxETDRS letters" to distinguish the scores from visual acuity measurements obtained using the ETDRS chart. It was assumed that one line equals five ETDRS points. The time in days to improvement of 2 or more lines is reported.
Time Frame: Baseline, Up to 17 Months
Population: All participants with improvement of 2 lines or more in BCVA.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | OZURDEX®
Number analyzed (Participants) | 27
days | 105.41 (184.50)

6. Secondary Outcome: Time to Improvement of 3 Lines or More in BCVA in the Study Eye
Description: BCVA following the injection of OZURDEX® is measured in the study eye using a special eye chart. BCVA measurements expressed in Snellen fractions were converted to logMAR units and approximate ETDRS letter scores based on the formula: approximate ETDRS letters = 85 + 50 x log10 (Snellen fraction). The converted scores hereinafter are referred to as "approxETDRS letters" to distinguish the scores from visual acuity measurements obtained using the ETDRS chart. It was assumed that one line equals five ETDRS points. The time in days to improvement of 3 or more lines is reported.
Time Frame: Baseline, Up to 17 Months
Population: All participants with improvement of 3 lines or more in BCVA.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | OZURDEX®
Number analyzed (Participants) | 23
days | 100.48 (172.84)

7. Secondary Outcome: Time to OZURDEX® Re-Injection in the Study Eye
Time Frame: Up to 17 Months
Population: All participants who had OZURDEX® re-injection.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | OZURDEX®
Number analyzed (Participants) | 7
days | 223.00 (54.71)

ADVERSE EVENTS:
Arm/Group | OZURDEX®
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 29/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OZURDEX® (N=43)
Increased intraocular pressure (Investigations) | 12
Ocular hypertension (Eye disorders) | 5
Conjunctival haemorrhage (Eye disorders) | 11
Chemosis (Eye disorders) | 4
Conjunctival hyperaemia (Eye disorders) | 10
Cortical/nuclear cataract (Eye disorders) | 4
Subcapsular cataract (Eye disorders) | 2
Vitreous floaters (Eye disorders) | 2
Eye pain (Eye disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.